CLINICAL TRIAL: NCT03865394
Title: Evaluation of the Safety and Efficacy of the Treatment of Chronic Wounds in Diabetic Foot Syndrome With the Use of Allogeneic Stem Cells Isolated From Adipose Tissue
Brief Title: Treatment of Chronic Wounds in Diabetic Foot Syndrome With Allogeneic Adipose Derived Mesenchymal Stem Cells
Acronym: 1ABC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Polish Stem Cells Bank S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1ABC Therapy; 267976/13/NCBR/2015 (Other Grant/Funding Number: The National Center for Research and Development, Poland); 2016-004109-15 (EudraCT Number); PL008125 (Other: EU tissue establishment code); Z4217 (Other: ISBT128 (Facility Identification Number))
Record Dates: First submitted 2018-11-08; First posted 2019-03-06 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: stromal vascular fraction; adipose-derived mesenchymal stem cells; chronic wounds; diabetes; foot ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic ADSC cells in fibrin solution (Experimental): Application of allogeneic ADSC stem cells in fibrin gel, to cover wound surface with thin cells layer.
  Therapy is based on standard procedure of diabetic foot ulcer treatment combined with application of allogeneic ADSC stem cells in fibrin solution onto the wound surface.
  Interventions: Biological: Application of allogeneic ADSC stem cells in fibrin gel
- Standard care in diabetic foot ulcer with aplication of fibrin gel to cover wound surface. (Active Comparator): Application of fibrin gel to cover wound surface.
  Interventions: Procedure: Standard care in diabetic foot ulcer

INTERVENTIONS:
Biological: Application of allogeneic ADSC stem cells in fibrin gel — Chronic wounds in diabetic foot ulcer will be covered with ADSC suspended in fibrin gel - single dose will be administered followed by weekly wound control.
  Arms: Allogeneic ADSC cells in fibrin solution
Procedure: Standard care in diabetic foot ulcer — Chronic wounds in diabetic foot ulcer will be covered with fibrin gel followed by weekly wound control.
  Arms: Standard care in diabetic foot ulcer with aplication of fibrin gel to cover wound surface.

SUMMARY:
The aim of this study is to investigate efficiency of applying of adipose-derived mesenchymal stem cells (ADSC) in treatment of chronic wounds in diabetic foot syndrome.

DETAILED DESCRIPTION:
The product will contain an active ingredient- human allogeneic adipose-derived mesenchymal stem cells (ADSC) cells suspended in the fibrin solution applied directly onto prepared wound bed, to form thin gel layer on the wound surface.

ELIGIBILITY:
Inclusion Criteria:

1. Signing informed consent form.
2. Above the age of 18
3. Voluntary participation in the research, following the requirements of the protocol and acceptance for procedures related with its implementation
4. Chronic wound in the course of diabetic foot syndrome, with the wound surface between 1 - 25 sq. cm, without evidence of active infection of the wound at the time of qualification to participate in the study
5. Blood level of glycated haemoglobin (HbA1c) <=11%
6. Satisfactory blood supply to the wound verified by the measurement of the oxygen level in the foot tissue (>=30 mmHg), or by the measurement of systolic blood pressure in posterior or anterior tibial artery (>=50 mmHg) of the affected limb.
7. General health condition, which according to the investigator's opinion, allows patient's participation in all study procedures.

Exclusion Criteria:

1. Lack of patient's cooperation
2. Wound etiology other than diabetic foot syndrome
3. Clinicaly significant limb ischemia as verified by the measurement of the oxygen level in the foot tissue (<30 mmHg), or by the measurement of systolic blood pressure in posterior or anterior tibial artery (<50 mmHg)
4. Active wound infection, which would require the treatment with antibiotics
5. Known allergy to ingredients of study product (thrombin, penicillin).
6. Active venous thromboembolism
7. Any systemic disease (acute or chronic) in the stage of exacerbation or not stabilized, that in the opinion of the investigator may hinder or make impossible a patient's participation in the study
8. Active cancer during chemotherapy or radiotherapy, or recent cancer, if the remission occured less than 5 years before joining the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in wound size | 8 weeks
  The comparison of the time required for the 50% reduction of initial wound size between patients in both study arms.
  The wound size changes will be assessed using digital 3D wound imaging medical device with image processing software, according to the following rules:
  * for wounds deeper than 0.5 cm - measurement of wound volume, or
  * for shallow wounds (less than 0.5 cm depth) - measurement of wound surface.

SECONDARY OUTCOMES:
Changes in wound morphology | 8 weeks
  Clinical assessment of wound morphology (and its changes during the treatment) in each treated patient, as well, as between patients in both study arms, expressed as:
  * the amount (1) and features (2) of wound exudate,
  * the presence of redness (3) and/or edema (4) in the wound surrounding skin,
  * the presence of granular tissue and fibrin (5) or epithelium (6) in the wound bed.
  The listed parameters will be assessed using simplified questionnaire adopted from Bates-Jensen Wound Assessment Tool (positions 7-13 from B-JWAT).
  Each of 6 abovementioned features will be assessed semiquantitatively using 1-5 points scale, (with "1" for a best state, and "5" for a worst state). The sum of points allocated to each parameter will be recorded as the wound score and used for further analysis.
  The healthy skin/healed wound should receive 6 points, whereas active wound, with exudate and inflammation will receive 30 points (the lower = the better / the higher = the worse).
Changes in pro-angiogenic factors expression | 8 weeks
  Evaluation of the expression (and its changes during the treatment) of selected pro-angiogenic factors, measured in wound biopsies.
  The changes will be analyzed for each tested individual separately, and compared between both study arms.
Changes in wound-associated pain | 8 weeks
  Evaluation of the wound-associated pain, assessed by the patient using visual analogue scale. The minimum value is 0 and means "no pain" and the maximum value is 10 and means "the worst possible pain". The lower value the better outcome.
  The changes will be analyzed for each tested individual separately, and compared between both study arms.
Changes in the quality of life | 8 weeks
  Evaluation of the patient's quality of life, assessed by the dedicated QoL questionnaire. The QoL questionnaire consists of 10 questions. Each question is scored 1 to 5. The minimum score is 10 and it means "the best possible state of health", and the maximum score is 50, which means ,,the worst possible state of health".
  The changes will be analyzed for each tested individual separately, and compared between both study arms.
Record of adverse events | 8 weeks
  Evaluation of the safety of ADSC application, assessed by the occurrence of any adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Beata Mrozikiewicz-Rakowska, . Assoc.Prof., Principal Investigator — Medical University of Warsaw, Department of Diabetology and Internal Diseases
Locations (1):
- Medical University of Warsaw, Department of Diabetology and Internal Diseases, Warsaw, Poland